CLINICAL TRIAL: NCT00764322
Title: Validating CYP2D6 Genotype-Guided Tamoxifen Therapy for a Multiracial U.S. Population
Brief Title: Studying Blood Samples From Women With Breast Cancer or Ductal Carcinoma In Situ Who Are Receiving Tamoxifen
Acronym: NRR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0801; P30CA016086 (NIH); 08-0483 (Other: UNC Biomedical IRB)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Menopausal Symptoms
Keywords: menopausal symptoms; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Tamoxifen; Gene Expression Profiling; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamoxifen 20 (Experimental): One arm, containing the ultra-rapid and extensive metabolizer genotypes, continues treatment with tamoxifen at 20mg.
  Interventions: Drug: tamoxifen citrate; Genetic: gene expression analysis; Other: pharmacogenomic studies; Other: questionnaire administration; Procedure: quality-of-life assessment
- Tamoxifen 40 (Active Comparator): This arm, containing the intermediate and poor metabolizer genotypes, receives escalated treatment with tamoxifen at 40mg.
  Interventions: Drug: tamoxifen citrate; Genetic: gene expression analysis; Other: pharmacogenomic studies; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: tamoxifen citrate — Women found to be IM or PM will undergo increased tamoxifen to 40 mg/day (20 mg bid). Drug is given orally on a daily basis.
  Other Names: Nolvadex; Soltamox
Genetic: gene expression analysis — Genetic analysis of blood sample.
Other: pharmacogenomic studies — Genetic analysis of blood sample.
Other: questionnaire administration — Questionnaire called the survey of participants. Questionnaires is self administered on paper documents and given pre-study, and at 4 months
Procedure: quality-of-life assessment — Self administration of a multiquestion questionnaire called the Functional Assessment of Cancer Therapy -Breast (FACT-B). Given pre-study, at 4 months and at 8-10 months.

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about differences in DNA and predict how well patients will respond to treatment and plan better treatment.

PURPOSE: This clinical trial is studying blood samples from women with breast cancer or ductal carcinoma in situ who are receiving tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the change in endoxifen levels after an increase in tamoxifen citrate dose from 20 mg to 40 mg in women with breast cancer or ductal breast carcinoma in situ with intermediate-metabolizing CYP2D6 genotypes.

Secondary

* To evaluate the tolerability of increasing the dose of tamoxifen citrate from 20 to 40 mg per day in these patients.
* To assess the feasibility of obtaining pharmacogenomic information from patients in the clinical setting and using it to guide changes in therapy.
* To examine CYP2D6 allele frequencies and endoxifen levels among African-American women taking tamoxifen citrate.
* To evaluate the change in plasma endoxifen levels after an increase in the tamoxifen citrate dose from 20 mg to 40 mg daily in patients with poor-metabolizing genotypes.
* To study patient understanding of pharmacogenomics and obstacles to participation in clinical trials based upon germline DNA.

OUTLINE: This is a multicenter study.

Blood samples are collected at baseline to determine CYP2D6 genotype and tamoxifen citrate metabolic status: poor-metabolizing (PM), intermediate-metabolizing (IM), or extensive-metabolizing (EM) alleles. Samples are also analyzed for plasma levels of endoxifen and N-desmethyltamoxifen and for endoxifen/N-desmethyltamoxifen ratio. Patients found to be IM or PM are notified to increased tamoxifen citrate to 40 mg/day for 4 months (in the absence of unacceptable toxicity) with repeat endoxifen and N-desmethyltamoxifen levels (and the ratio) at the end of this time.

All patients complete Quality Of Life (QOL) and Menopausal Symptoms Scale (MSS) questionnaires at baseline and after 4 months of treatment. Toxicities are assessed at the end of 4 months. Patients undergo repeat questionnaire assessment of their understanding of the use of pharmacogenomics in clinical decision-making. Some patients also undergo a 30-minute, baseline interview regarding attitudes and experience towards participation in a pharmacogenomics study.

Patients who choose to be informed of the results of their genotyping are contacted by letter, along with their physicians, and offered genetic counseling to discuss the significance of these results.

After completion of study therapy, patients are followed at 3-6 months, including toxicity assessment and QOL and MSS questionnaires.

ELIGIBILITY:
Inclusion:

Histologically confirmed invasive carcinoma of the breast or ductal breast carcinoma in situ Has been receiving tamoxifen citrate at a dose of 20 mg/day for at least 4 months either for the treatment of invasive or non-invasive carcinoma of the breast or for breast cancer recurrence prevention

* Expected duration of tamoxifen citrate treatment at least 6 months Hormone receptor status not specified Concurrent participation in non-treatment studies allowed provided it will not interfere with participation in this study Menopausal status not specified Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Life expectancy ≥ 6 months Absolute Neutrophil Count (ANC) ≥ 1.0 x 10^9/L Platelet count ≥ 100 x 10^9/L Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times Upper Limit of Normal (ULN) Total bilirubin ≤ 2.5 times ULN Creatinine clearance ≥ 50 mL/min Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No limitations to number of prior therapies
* No limitations for prior radiotherapy
* More than 14 days since prior and no other concurrent investigational agent

Exclusion:

Not pregnant or nursing No active, serious infection or medical or psychiatric illness likely to preclude study participation No psychiatric conditions that would preclude study compliance or informed consent No history of venous thromboembolism, transient ischemic attack, or cerebral vascular accident No history of allergic reaction to tamoxifen citrate or any of its reagents No concurrent coumadin

No concurrent medications known to inhibit CYP2D6, including any of the following:

* Amiodarone
* Haloperidol
* Indinavir
* Ritonavir
* Quinidine

No concurrent selective serotonin reuptake inhibitors, except the following:

* Venlafaxine
* Citalopram

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2008-06-18; Primary Completion 2010-09-28 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; William J. Irvin, MD, Principal Investigator — Bon Secours Virginia Health System / Bon Secours Cancer Institute
Locations (7):
- United States (7):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00764322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from breast cancer patients at Lineberger Comprehensive Cancer Center who had received tamoxifen for at least 4 months.
Pre-assignment Details: One patient was a screen failure
Period: Overall Study
Arm/Group | Patients Enrolled
Started | 500
Completed | 480
Not Completed | 20
Not completed — Withdrawal by Subject | 11
Not completed — No CYP2D6 genotyping | 9

BASELINE CHARACTERISTICS:
Groups:
- Extensive and Ultra-rapid Metabolizers: Those with the highest endoxifen concentrations as measured at baseline.
- Intermediate and Poor Metabolizers: Genotype-guided escalation of the tamoxifen dose from 20mg to 40mg/day.
- Total: Total of all reporting groups
Arm/Group | Extensive and Ultra-rapid Metabolizers | Intermediate and Poor Metabolizers | Total
Number analyzed (Participants) | 161 | 319 | 480
Age, Continuous [Median (Full Range); unit: years]
  Median | 51 [30 to 95] | 50 [25 to 88] | 50 [25 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 319 | 480
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 61 | 74
  White | 140 | 250 | 390
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 319 | 480
Menopausal status [Count of Participants; unit: Participants]
  Pre/peri- | 70 | 154 | 224
  Post- | 91 | 165 | 256
Duration of Tamoxifen treatment (years) [Median (Full Range); unit: years] | 0.88 [0.31 to 9.69] | 0.98 [0.28 to 15.86] | 0.93 [0.28 to 15.86]
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 92 | 169 | 261
  No | 69 | 150 | 219
Tamoxifen indication [Count of Participants; unit: Participants] — Population: One patient could not be included because indication was not supplied.
  Participants
    number analyzed (Participants) | 161 | 318 | 479
    Invasive Disease | 144 | 263 | 407
    DCIS | 17 | 49 | 66
    Other | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Endoxifen Concentrations in Participants Receiving Tamoxifen Citrate Dose of 20 mg or 40 mg Stratified by the Metabolizing CYP2D6 Genotypes
Description: Measurements of plasma concentrations of the key active metabolite of tamoxifen, endoxifen, were measured at baseline and after 4 months of treatment; The most common CYP2D6 alleles have been grouped by functional activity classifications with descending activity: ultra-rapid (UM), extensive (EM), intermediate (IM) or poor (PM) metabolism. A given patient has two alleles, giving them 10 possible allelic combinations, or diplotypes (UM/UM, UM/EM, EM/EM, etc.). These diplotypes are collapsed into four phenotypes, UM, EM, IM or PM.
Time Frame: 4 months
Population: Baseline measurements are reported on all 353 subjects, while the 4 month levels are reported only for patients who completed 4 months of treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ultra-rapid Metabolizers: Those with the highest transformation of the CYP2D6 genotype to allelic activity
- Extensive Metabolizers: Those with the most normal transformation of the CYP2D6 genotype to allelic activity
- Intermediate Metabolizers: Those with reduced transformation of the CYP2D6 genotype to allelic activity Genotype-guided escalation of the tamoxifen dose from 20mg to 40mg/day.
- Poor Metabolizers: Those with no transformation of the CYP2D6 genotype to allelic activity Genotype-guided escalation of the tamoxifen dose from 20mg to 40mg/day.
Arm/Group | Ultra-rapid Metabolizers | Extensive Metabolizers | Intermediate Metabolizers | Poor Metabolizers
Number analyzed (Participants) | 5 | 119 | 212 | 17
ng/mL
  Baseline endoxifen concentration | 8.4 (4.59) | 10.00 (6.00) | 7.10 (4.77) | 3.42 (2.75)
  4-Month endoxifen concentration: number analyzed (Participants) | 4 | 106 | 179 | 13
  4-Month endoxifen concentration | 15.35 (5.48) | 9.30 (5.03) | 10.74 (7.36) | 5.52 (2.57)

2. Secondary Outcome: Number of Participants With Pulmonary Embolism (PE), Deep Vein Thrombosis (DVT), Stroke, and/or Endometrial Cancer
Description: The doubling of tamoxifen dose is defined as "unacceptable" (i.e., not tolerable) if the prevalence of Pulmonary embolism (PE), Deep vein thrombosis (DVT), stroke, or endometrial cancer, either individually or in any combination, is greater than 2%.
Time Frame: Approximately ten months from registration to last follow-up
Population: Incidence of unacceptable adverse events among all patients who completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Tamoxifen 20 | Tamoxifen 40
Number analyzed (Participants) | 161 | 319
Participants
  Pulmonary embolism (PE) | 0 | 0
  Deep vein thrombosis (DVT) | 0 | 0
  Stroke | 0 | 0
  Endometrial cancer | 0 | 0

3. Secondary Outcome: Change in Median Endoxifen Concentrations to Determine Feasibility of Obtaining Pharmacogenomic Information From Patients in the Clinical Setting and Using it to Guide Changes in Therapy
Description: If the key active tamoxifen metabolite, endoxifen, could be significantly increased by genotype-guided tamoxifen dosing in patients with intermediate CYP2D6 metabolism (by increasing tamoxifen dosing based on CYP2D6 genotype), then the study would be deemed feasible and the accrual expanded.
Time Frame: Baseline and 4 months after dose increase
Population: This was based on the initial 119 subjects enrolled (based on initial sample size of 100) and of those, the 89 that completed 4 months of tamoxifen therapy
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Extensive Metabolizers: Those with the highest endoxifen concentrations as measured at baseline.
- Intermediate Metabolizers; Poor Metabolizers: Genotype-guided escalation of the tamoxifen dose from 20mg to 40mg/day.
Arm/Group | Extensive Metabolizers | Intermediate Metabolizers | Poor Metabolizers
Number analyzed (Participants) | 29 | 51 | 9
ng/mL | -1.5 [-28 to 11.2] | 7.6 [-0.6 to 23.9] | 6.1 [2.6 to 12.5]

4. Secondary Outcome: CYP2D6 Allele Frequencies and Endoxifen Levels Among African-American Women Taking Tamoxifen Citrate
Description: Mean endoxifen levels by CYP2D6 genotype among African Americans. Measurements of plasma concentrations of the key active metabolite of tamoxifen, endoxifen, were measured at baseline.The most common CYP2D6 alleles have been grouped by functional activity classifications with descending activity: ultra-rapid (UM), extensive (EM), intermediate (IM) or poor (PM) metabolism. A given patient has two alleles, giving them 10 possible allelic combinations, or diplotypes (UM/UM, UM/EM, EM/EM, etc.). These diplotypes are collapsed into four phenotypes, UM, EM, IM or PM.
Time Frame: baseline
Population: Only participants who self-identified as African American were included in this analysis
Measure: Mean (Full Range); unit: ng/ml
Groups:
- African Americans: Participants who self identified as African American Race
Arm/Group | African Americans
Number analyzed (Participants) | 52
ng/ml
  UM: number analyzed (Participants) | 1
  UM | 14.58 [14.58 to 14.58]
  EM: number analyzed (Participants) | 8
  EM | 9.69 [1.08 to 21.98]
  IM: number analyzed (Participants) | 42
  IM | 7.09 [1.07 to 20.89]
  PM: number analyzed (Participants) | 1
  PM | 0.8 [0.8 to 0.8]

5. Secondary Outcome: Change in Plasma Endoxifen Levels After an Increase in Tamoxifen Citrate Dose From 20 mg to 40 mg Daily in Patients With Poor-metabolizing Genotypes
Description: The intrapatient change in median endoxifen levels were calculated between baseline and 4 months after the increase in dose of Tamoxifen from 20mg/day to 40 mg/day
Time Frame: Baseline and 4 months after dose increase
Population: Analysis limited to only those subjects with the Poor Metabolizing (PM) genotype who were evaluable at baseline
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Poor Metabolizers
Number analyzed (Participants) | 11
ng/mL | 6.1 [2.6 to 12.5]

6. Secondary Outcome: Patient Understanding of Pharmacogenomics
Description: To examine patients' beliefs about how hypothetical genotype information would affect their perceived recurrence risk and benefits of tamoxifen therapy, participants were given experimentally manipulated 6 vignettes to describe hypothetical tamoxifen treatment (no or yes) and hypothetical genotype (EM, IM or PM). For each vignette, participants gave their perceived recurrence risk (RR; 0-100%)
Time Frame: baseline
Population: Of 377 patients who were eligible to complete the survey, 320 patients completed the survey and 57 returned incomplete surveys
Measure: Mean (Full Range); unit: percent chance of recurrence
Groups:
- All Participants: All participants in the main study who consented to this additional survey
Arm/Group | All Participants
Number analyzed (Participants) | 320
percent chance of recurrence
  Perceived RR -No tamoxifen/EM | 47 [0 to 100]
  Perceived RR -No tamoxifen/iM | 48 [0 to 100]
  Perceived RR -No tamoxifen/PM | 53 [0 to 100]
  Perceived RR - tamoxifen/EM | 22 [0 to 100]
  Perceived RR -tamoxifen/IM | 30 [0 to 100]
  Perceived RR -tamoxifen/PM | 40 [0 to 100]

ADVERSE EVENTS:
Time Frame: Approximately ten months from on-study to last follow-up visit
Groups:
- Ultra-rapid and Extensive Metabolizers: Those with the highest endoxifen concentrations as measured at baseline.
Arm/Group | Ultra-rapid and Extensive Metabolizers | Intermediate Metabolizers | Poor Metabolizers
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/290 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/161 | 3/290 | 0/29
Other Adverse Events (participants affected / at risk) | 149/161 | 274/290 | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultra-rapid and Extensive Metabolizers (N=161) | Intermediate Metabolizers (N=290) | Poor Metabolizers (N=29)
Hemorrhage, GU (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Mood alteration (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Depression
thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — thrombosis, vascular access related
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultra-rapid and Extensive Metabolizers (N=161) | Intermediate Metabolizers (N=290) | Poor Metabolizers (N=29)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 | 11 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 | 3 | 0
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 5 | 3 | 0
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 4 | 6 | 0
Cataract (Eye disorders) | 3 | 8 | 0
Cognitive disturbance (Nervous system disorders) | 13 | 27 | 3
Constipation (Gastrointestinal disorders) | 8 | 18 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 9 | 2
Distension/bloating, abdominal (Gastrointestinal disorders) | 5 | 9 | 0
Dizziness (Nervous system disorders) | 5 | 14 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 0
Edema: limb (General disorders) | 10 | 19 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 42 | 64 | 5
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2 | 6 | 0 — Verbatim: Mouth problems; dry mouth; dysphagia with regurgitation, requiring dilation; gastroparesis; taste alteration; anorexia; gastric dumping syndrome; teeth sensitivities
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 8 | 17 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 5 | 10 | 0
Hemorrhage, GU - Vagina (Blood and lymphatic system disorders) | 0 | 4 | 2
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 3 | 2 | 0 — Verbatim: Blood flecking in stools; epistaxis; hematemisis; nose hemorrhage; bloodshot eyes
Hemorrhoids (Gastrointestinal disorders) | 2 | 4 | 0
Hot flashes/flushes (Vascular disorders) | 124 | 230 | 23
Hypertension (Vascular disorders) | 3 | 11 | 0
Incontinence, urinary (Renal and urinary disorders) | 13 | 28 | 3
Infection with unknown ANC (Infections and infestations) | 0 | 9 | 0
Insomnia (Psychiatric disorders) | 26 | 42 | 4
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 9 | 14 | 0
Joint - Function (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0
Libido (Reproductive system and breast disorders) | 16 | 24 | 3
Lymphedema-related fibrosis (Vascular disorders) | 0 | 5 | 0
Memory impairment (Nervous system disorders) | 6 | 16 | 0
Mood alteration (Psychiatric disorders) | 2 | 4 | 0
Mood alteration - Agitation (Psychiatric disorders) | 5 | 9 | 4
Mood alteration - Anxiety (Psychiatric disorders) | 20 | 17 | 0
Mood alteration - Depression (Psychiatric disorders) | 14 | 13 | 2
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 5 | 11 | 0 — Verbatim: broken wrist; feet stiff; weakness; avascular necrosis; leg cramps; difficulty walking; fractured vertebrae; joint difficulties right thumb; osteopenia; pulled back; rotator cuff tear; tennis elbow; fractured elbow; stiffness
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 7 | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 6 | 18 | 0
Neurology - Other (Specify, __) (Nervous system disorders) | 0 | 7 | 0 — Verbatim: hallucinations at night; seizures; felt drunk; claustrophobia; feeling weird; handwriting worsened, near syncope
Neuropathy- sensory (Nervous system disorders) | 15 | 22 | 0
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 | 6 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 15 | 28 | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 4 | 11 | 0
Pain - Breast (Musculoskeletal and connective tissue disorders) | 13 | 22 | 0
Pain - Buttock (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pain - Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 16 | 14 | 3
Pain - Head/headache (Nervous system disorders) | 15 | 42 | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 40 | 58 | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 15 | 38 | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Pain - Other (Specify, __) (General disorders) | 4 | 6 | 0
Palpitations (Cardiac disorders) | 4 | 5 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 6 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 | 6 | 2
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 9 | 17 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 6 | 12 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 2 | 0
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 20 | 44 | 2
Vaginal dryness (Reproductive system and breast disorders) | 32 | 66 | 8
Vaginitis (Reproductive system and breast disorders) | 3 | 3 | 0
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 | 4 | 0
Vision-blurred vision (Eye disorders) | 8 | 21 | 0
Weight gain (Investigations) | 14 | 33 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No